CLINICAL TRIAL: NCT02845817
Title: Requests for Euthanasia and Assisted Suicide: a Prospective, Multicenter and Qualitative Study of Their Frequency and Characteristics, of Patients' Motivations and Their Evolution
Brief Title: Requests for Euthanasia and Assisted Suicide
Acronym: DESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Maison Médicale Jeanne Garnier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DESA
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Palliative Care; End of Life; Euthanasia; Assisted Suicide; Qualitative Research
MeSH Terms: conditions — Death; Suicide, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Qualitative research (Other): Semi-structured interviews
  Interventions: Other: Qualitative research

INTERVENTIONS:
Other: Qualitative research — Semi-structured interviews

SUMMARY:
This study take place in the palliative care units of Burgundy-Franche-Comté regions and at the Maison Médicale Jeanne Garnier. The main aim of this project is to analyze and understand the meaning of explicit requests to hasten death (euthanasia and assisted suicide).

This involves conducting interviews with patients, carers to whom the request has been expressed and a relative chosen by the patient. This study aims to describe the request over time. This will be done through two series of interviews, one as soon as it is first expressed, then one week later.

ELIGIBILITY:
Inclusion Criteria:

* Adult not under guardianship or curatorship,
* Hospitalized in palliative care units of Bourgogne-Franche-Comté region and in the Maison Médicale Jeanne Garnier in Paris,
* At the end of life due to advanced stage disease or a major change in the state of health of an elderly person,
* They have made an explicit request for euthanasia or assisted suicide,
* They are in capacity to meet researchers for interview,
* Having consented to interviews,
* They are covered by the French social security system.

Exclusion Criteria:

* Adult under guardianship or curatorship,
* They are underage,
* They are not hospitalized in Palliative Care Unit of Bourgogne-Franche-Comté region and in the Maison Médicale Jeanne Garnier,
* The request was expressed by another person or not explicit,
* They didn't consent to interviews,
* The request appears in the context of a situation other than illness or a general change in state of health
* They are not in capacity to meet researchers for interviews.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
70 semi-structured interviews | 12 months
  Qualitative data analysis - Theoretical concept saturation and thematic analyses. [analyze and understand the meaning of explicit requests to hasten death (euthanasia and assisted suicide)]

CONTACTS AND LOCATIONS:
Overall Officials: Régis AUBRY, PR, Principal Investigator — Centre Hospitalier Universitaire de Besançon; Danièle LEBOUL, MCU, Principal Investigator — Maison Médicale Jeanne Garnier; Frédéric GUIRIMAND, DR, Principal Investigator — Maison Médicale Jeanne Garnier; Aline CHASSAGNE, IRC, Principal Investigator — Centre Hospitalier Universitaire de Besançon; Florence MATHIEU-NICOT, Phd, Principal Investigator — Centre Hospitalier Universitaire de Besançon; Anne BOUSQUET, Phd, Principal Investigator — Maison Médicale Jeanne Garnier
Locations (1):
- CHRU Besançon - Palliative Care Unit, Besançon, Bourgogne-Franche-Comté, France